CLINICAL TRIAL: NCT02134015
Title: Phase 3, Randomized, Placebo-Controlled, Double-Blind, Multi-Center, Two-Part Study of Patritumab (U3-1287) In Combination With Erlotinib in EGFR Wild-type Subjects With Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) Who Have Progressed on at Least One Prior Systemic Therapy
Brief Title: Study of Patritumab in Combination With Erlotinib in Subjects With Locally Advanced or Metastatic Non-Small-Cell Lung Cancer (NSCLC). (HER3-Lung)
Acronym: HER3-Lung
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Pre-defined criteria for continuation were not reached
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U31287-A-U301; 2013-004371-12 (EudraCT Number)
Record Dates: First submitted 2014-04-08; First posted 2014-05-08 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Lung Cancer; Non-small Cell Lung Cancer
Keywords: Carcinoma; Non-Small-Cell Lung; Lung Neoplasms; Bronchogenic; Bronchial Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Erlotinib; Therapeutic Uses; Pharmacologic Actions; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma; Bronchial Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases | interventions — patritumab; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo + erlotinib (Experimental): Placebo infusion every 3 weeks and oral erlotinib 150 mg/day
  Interventions: Drug: Erlotinib; Drug: Placebo
- Patritumab + erlotinib (Experimental): Infusion of Patritumab (loading dose of 18 mg/kg, followed by 9 mg/kg every 3 weeks) and oral erlotinib 150 mg/day
  Interventions: Drug: Patritumab; Drug: Erlotinib

INTERVENTIONS:
Drug: Patritumab — Infusion of Patritumab (loading dose of 18 mg/kg, followed by 9 mg/kg every 3 weeks)
  Other Names: U3-1287
  Arms: Patritumab + erlotinib
Drug: Erlotinib — Oral erlotinib 150 mg/day
Drug: Placebo — Placebo infusion every 3 weeks
  Other Names: Matching Placebo
  Arms: Placebo + erlotinib

SUMMARY:
1. Part A: Subjects will receive Patritumab or placebo with erlotinib. Progression-free survival will be the primary outcome. Subjects will need to have Epidermal Growth Factor Receptor (EGFR) wild-type, locally advance or metastatic NSCLC and have their cancer progressed after at least one prior systemic anti-cancer therapy, available recent or archival tumor specimen and may not have had previous EGFR-targeted regimen, anti-HER2 (Human Epidermal Growth Factor Receptor 2), anti-HER3, or anti-HER4 therapy. Subjects may have high heregulin or low heregulin.
2. Part B: Subjects will receive Patritumab or placebo with erlotinib. Overall survival will be the primary outcome. Subjects will need to have EGFR wild-type, locally advance or metastatic NSCLC and have their cancer progressed after at least one prior systemic anti-cancer therapy, available recent or archival tumor specimen and may not have had previous EGFR-targeted regimen, anti-HER2, anti-HER3, or anti-HER4 therapy. Only subjects with high heregulin will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Must be greater or equal to 20 years of age
2. Must have cytologically or histologically confirmed NSCLC with either:

   * Metastatic disease (Stage IV) OR
   * Stage IIIB disease not amenable to surgery or curative intent.

   Note: It is permissible to use either AJCC Version 6.0 or the AJCC Version 7.0 staging system. For sites that use AJCC Version 7.0, T4M0 patients with other ipsilateral nodules and N0-N2 are still eligible.
3. If tumor histology is adenocarcinoma, must have wild-type EGFR genotype as assessed by a validated assay that includes exon 19 deletion and exon 21 (L858R) substitution.
4. Must have received one or two prior lines of systemic chemotherapy for advanced or metastatic disease, one of which must be a platinum-doublet therapy.
5. Must have disease progression or recurrence documented by radiographic assessment following treatment after last chemotherapy or chemoradiation regimen (completed within the previous 12 months).
6. Must have available recent (before treatment start) or archival tumor specimen.
7. Must have measurable disease for Part A, measurable disease or non-measurable disease for Part B
8. Must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
9. Must have adequate hematological function
10. Must have adequate renal function
11. Must have adequate hepatic function
12. Agreement to use effective contraception while on treatment and for at least 6 months after end of treatment
13. Must have provided informed consent for study participation.

Exclusion Criteria:

1. Lung adenocarcinoma with an Anaplastic Lymphoma Kinase (ALK) gene rearrangement
2. Left ventricular ejection fraction (LVEF) less than 45%
3. Prior EGFR-targeted regimen, anti-HER2, anti-HER3, or anti-HER4 therapy
4. History of other malignancies, except adequately treated non-melanoma skin cancer, curatively treated in-situ disease, or other solid tumors curatively treated with no evidence of disease for greater or equal to 5 years
5. History of corneal disease
6. History of interstitial lung disease (ILD)
7. Clinically active brain metastases
8. Uncontrolled hypertension
9. Clinically significant ECG changes
10. Clinically significant (in the opinion of the Investigator) ascites or pleural effusion requiring chronic medical intervention
11. Myocardial infarction within 1 year before enrollment, symptomatic congestive heart failure, unstable angina, or unstable cardiac arrhythmia requiring medication
12. Treatment with anticancer therapy, antibody-based therapy, retinoid therapy, or hormonal therapy within 4 weeks before study drug treatment
13. Therapeutic radiation therapy or major surgery within 4 weeks before study drug treatment; or palliative radiation within 2 weeks before study drug treatment
14. Participation in clinical drug trials within 4 weeks
15. Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals, known human immunodeficiency virus (HIV) infection, or active hepatitis B or C infection.
16. History of hypersensitivity to any of the study drugs or to any excipients.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2014-03; Primary Completion 2016-11-11 (Actual); Study Completion 2016-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (98):
- United States (26):
  - Glendale, Arizona
  - Duarte, California
  - La Verne, California
  - Los Angeles, California
  - San Francisco, California
  - Port Saint Lucie, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Maywood, Illinois
  - Goshen, Indiana
  - Louisville, Kentucky
  - Grand Rapids, Michigan
  - Saint Cloud, Minnesota
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Columbus, Ohio
  - Bend, Oregon
  - Portland, Oregon
  - Redmond, Oregon
  - Chattanooga, Tennessee
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Salt Lake City, Utah
  - Arlington, Virginia
  - Seattle, Washington
- Belgium (7):
  - Brasschaat, Antwerpen
  - Brussels, Brussels Capital
  - Charleroi, Hainaut
  - Charleroi
  - Ghent
  - Liège
  - Yvoir
- Canada (5):
  - Hamilton, Ontario
  - Kingston, Ontario
  - Toronto, Ontario
  - Lévis, Quebec
  - Montreal, Quebec
- Czechia (2):
  - Ostava-Poruba
  - Ostrava-Poruba
- Germany (15):
  - Esslingen am Neckar, Baden-Wurttemberg
  - Gerlingen, Baden-Wurttemberg
  - Heidelberg, Baden-Wurttemberg
  - Ulm, Baden-Wurttemberg
  - Villingen-Schwenningen, Baden-Wurttemberg
  - Gauting, Bavaria
  - Munich, Bavaria
  - Frankfurt am Main, Hesse
  - Immenhausen, Hesse
  - Cologne, North Rhine-Westphalia
  - Rheine, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Halle, Saxony-Anhalt
  - Großhansdorf, Schleswig-Holstein
  - Giessen
- Hungary (4):
  - Székesfehérvár, Fejér
  - Győr, Győr-Moson-Sopron
  - Szolnok, Jász-Nagykun-Szolnok
  - Tatabánya
- Italy (15):
  - Meldola, Forli
  - Sora, Frosinone
  - Lecco, Lombardy
  - Benevento
  - Bologna
  - Cremona
  - Faenza
  - Genova
  - Milan
  - Napoli
  - Perugia
  - Ravenna
  - Rimini
  - Roma
  - Rozzano
- Poland (7):
  - Torun, Kuyavian-Pomeranian Voivodeship
  - Otwock, Masovian Voivodeship
  - Gdansk, Pomeranian Voivodeship
  - Szczecin, West Pomeranian Voivodeship
  - Krakow
  - Prabuty
  - Warsaw
- Spain (11):
  - A Coruña, A Coruña
  - Seville, Andalusia
  - Valencia, Valenciana, Comunidad
  - Alicante
  - Barcelona
  - Burgos
  - Madrid
  - Manresa
  - Palma de Mallorca
  - Valencia
  - Zaragoza
- United Kingdom (6):
  - Stevenage, Hertfordshire
  - London
  - Metropolitan Borough of Wirral
  - Northwood
  - Rickmansworth
  - Southampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was randomized on 11 Jun 2014, and the last patient's last visit occurred on 11 Nov 2016. All randomized participants received study treatment and were included in both the Full Analysis Set and the Safety Analysis Set.
Pre-assignment Details: Of 537 patients screened, a total of 145 patients were randomized into this trial in 9 countries: United States (26 at 12 sites), Spain (19 at 5 sites), Hungary (18 at 4 sites), Italy (20 at 6 sites), Great Britain (11 at 5 sites), Poland (30 at 3 sites), Germany (16 at 6 sites), Canada (2 at 1 site) and Belgium (3 at 1 site).
Period: Overall Study
Arm/Group | Placebo + Erlotinib | Patritumab + Erlotinib
Started | 71 | 74
Completed | 0 | 0
Not Completed | 71 | 74
Not completed — Protocol Violation | 0 | 1
Not completed — Death | 2 | 1
Not completed — Reason not provided | 1 | 2
Not completed — Clinical progression | 14 | 7
Not completed — Progressive disease (per RECIST 1.1) | 40 | 43
Not completed — Study terminated by sponsor | 2 | 3
Not completed — Adverse Event | 9 | 10
Not completed — Withdrawal by Subject | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Erlotinib | Patritumab + Erlotinib | Total
Number analyzed (Participants) | 71 | 74 | 145
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 40 | 78
  >=65 years | 33 | 34 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (9.15) | 63.9 (8.25) | 63.6 (8.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 30 | 52
  Male | 49 | 44 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 59 | 66 | 125
  Unknown or Not Reported | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 71 | 70 | 141
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Histology subtype [Count of Participants; unit: Participants]
  Adenocarcinoma | 39 | 40 | 79
  Squamous | 28 | 28 | 56
  Large Cell | 1 | 1 | 2
  Other | 3 | 5 | 8
Histology subtype (for randomization) [Count of Participants; unit: Participants]
  Adenocarcinoma | 38 | 40 | 78
  Squamous-cell carcinoma/Not otherwise specified | 33 | 34 | 67
Eastern Cooperative Oncology Group (ECOG) Score [Count of Participants; unit: Participants]
  0 - Fully Active | 24 | 25 | 49
  1 - Restricted in Physically Strenuous Activity | 47 | 49 | 96
Heregulin (HRG) expression from Interactive Web/Voice Response System (IXRS) [Count of Participants; unit: Participants]
  HRG High | 48 | 47 | 95
  HRG Low | 23 | 27 | 50

OUTCOME MEASURES:

1. Primary Outcome: Part A: Progression Free Survival (PFS) in Heregulin-high Participants
Description: PFS is defined as the time from the date of randomization to the earlier of the dates of first objective documentation of radiographic disease progression (as per RECIST Version 1.1 per investigator assessment) or death resulting from any cause.
  Kaplan-Meier Estimate. Confidence interval (CI) for median was computed using the Brookmeyer-Crowley method. 80% confidence interval is included in the data table.
Time Frame: by trial termination (at 20 months)
Measure: Number (80% Confidence Interval); unit: months
Arm/Group | Placebo + Erlotinib | Patritumab + Erlotinib
Number analyzed (Participants) | 48 | 47
months | 2.7 [1.7 to 2.9] | 1.9 [1.4 to 3.5]

2. Primary Outcome: Part A: Progression Free Survival (PFS) in Heregulin-low Participants
Description: as for outcome 1
Time Frame: by trial termination (at 20 months)
Measure: Number (80% Confidence Interval); unit: months
Arm/Group | Placebo + Erlotinib | Patritumab + Erlotinib
Number analyzed (Participants) | 23 | 27
months | 2.8 [1.4 to 4.2] | 1.5 [1.4 to 2.7]

3. Primary Outcome: Part B: Overall Survival
Description: Percentage of participants still alive at the end of Part B
Time Frame: 4 years
Population: No participants were analyzed for Part B endpoints because the trial was terminated at the end of Part A.
Arm/Group | Placebo + Erlotinib | Patritumab + Erlotinib
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Part A: Overall Survival in HRG High Participants
Description: Key secondary efficacy endpoint: Percentage of participants who survived for the length of the trial
Time Frame: by trial termination (at 20 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Erlotinib | Patritumab + Erlotinib
Number analyzed (Participants) | 48 | 47
Participants | 15 | 17

5. Secondary Outcome: Part A: Key Secondary Efficacy Endpoint: Overall Survival in HRG Low Participants
Description: Key secondary efficacy endpoint: Percentage of participants who survived for the length of the trial
Time Frame: by trial termination (at 20 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Erlotinib | Patritumab + Erlotinib
Number analyzed (Participants) | 23 | 27
Participants | 7 | 8

6. Secondary Outcome: Part B: Key Secondary Efficacy Endpoint: PFS, TTD
Description: PFS is defined as the time from the date of randomization to the earlier of the dates of first objective documentation of radiographic disease progression (TTD, as per RECIST Version 1.1 per investigator assessment) or death resulting from any cause.
Time Frame: 4 years
Population: No participants were analyzed for Part B endpoints because the trial was terminated at the end of Part A.
Arm/Group | Placebo + Erlotinib | Patritumab + Erlotinib
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Part A: Objective Response Rate (ORR) in HRG High Participants
Description: Key secondary efficacy endpoint: Objective response is defined as percentage of participants achieving complete response (CR) or partial response (PR)
  Denominator for percentages is the number of subjects with measurable disease in the full analysis set. The best overall response is the best response [in the order of CR, PR, stable disease (SD), and progressive disease (PD)] among all overall responses recorded from the start of treatment until the subject withdraws from the study. If there is no post-baseline tumor assessment or all post-baseline tumor assessments with overall response being Inevaluable captured in the CRF, the best overall response is classified as Inevaluable.
Time Frame: by trial termination (at 20 months)
Population: Evaluable participants in the full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Erlotinib | Patritumab + Erlotinib
Number analyzed (Participants) | 48 | 46
Participants | 3 | 1

8. Secondary Outcome: Part A: Objective Response Rate (ORR) in HRG Low Participants
Description: Key secondary efficacy endpoint: Objective response is defined as percentage of participants achieving complete response or partial response
  Denominator for percentages is the number of subjects with measurable disease in the full analysis set. The best overall response is the best response (in the order of CR, PR, SD, and PD) among all overall responses recorded from the start of treatment until the subject withdraws from the study. If there is no post-baseline tumor assessment or all post-baseline tumor assessments with overall response being Inevaluable captured in the CRF, the best overall response is classified as Inevaluable.
Time Frame: by trial termination (at 20 months)
Population: Evaluable participants in the full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Erlotinib | Patritumab + Erlotinib
Number analyzed (Participants) | 22 | 27
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: 53 days after the last dose of patritumab/placebo or 30 days after the last dose of erlotinib, whichever is later (within the length of the trial, which was 2 years, 7 months)
Description: Treatment emergent (TE) adverse events (AEs) are reported for patritumab only. If relatedness is missing, the AE is counted as related to patritumab.
Arm/Group | Placebo + Erlotinib | Patritumab + Erlotinib
All-Cause Mortality (participants affected / at risk) | 5/71 | 5/74
Serious Adverse Events (participants affected / at risk) | 29/71 | 27/74
Other Adverse Events (participants affected / at risk) | 66/71 | 68/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Erlotinib (N=71) | Patritumab + Erlotinib (N=74)
Deep vein thrombosis (Vascular disorders) | 1 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
General physical health deterioration (General disorders) | 1 | 2
Asthenia (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Aphagia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Swollen tongue (Gastrointestinal disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 1
Bronchitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Erlotinib (N=71) | Patritumab + Erlotinib (N=74)
Pruritus (Vascular disorders) | 4 (6) | 6 (7)
Weight decreased (Investigations) | 8 (9) | 10 (11)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 6 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (21) | 9 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 10 (14)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 5 (7)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Dizziness (Nervous system disorders) | 5 (5) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (3) | 4 (4)
Fatigue (General disorders) | 17 (23) | 11 (12)
Oedema peripheral (General disorders) | 6 (6) | 5 (5)
Asthenia (General disorders) | 5 (6) | 5 (5)
Chest pain (General disorders) | 4 (5) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 22 (41) | 39 (62)
Nausea (Gastrointestinal disorders) | 16 (18) | 15 (19)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 11 (18)
Vomiting (Gastrointestinal disorders) | 7 (8) | 10 (13)
Constipation (Gastrointestinal disorders) | 2 (2) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 5 (7)
Rash (Skin and subcutaneous tissue disorders) | 26 (46) | 28 (57)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 6 (7) | 13 (23)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (7) | 13 (14)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (4) | 6 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (5)
Decreased appetite (Metabolism and nutrition disorders) | 13 (16) | 17 (21)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (7) | 7 (17)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Paronychia (Infections and infestations) | 3 (4) | 7 (16)
Rhinitis (Infections and infestations) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes